CLINICAL TRIAL: NCT03293030
Title: Immunogenetic Profiling of Dupilumab for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dupilumab Immunogenetics
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema; Eczema; Atopic Dermatitis and Related Conditions
Keywords: atopic dermatitis; eczema; dupilumab; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupilumab treatment (Experimental): 15 subjects will receive dupilumab for a treatment period of 52 weeks (i.e. last injection on week 50). All subjects will undergo skin biopsies for molecular profiling.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab treatment
  Other Names: Dupixent

SUMMARY:
This is a single-arm, open-label study to examine the effect of dupilumab on the immunologic and genetic environment within atopic dermatitis skin lesions.

DETAILED DESCRIPTION:
Fifteen subjects with moderate to severe AD will receive dupilumab for a treatment period of 52 weeks (i.e. last injection on week 50). Biopsy samples from AD subjects and surgical discard samples will undergo molecular profiling. Skin swabs and stool samples will be collected and banked for future analysis. The reason to treat patients for 52 weeks is to have the ability to correlate early molecular events with clinical outcomes at week 52.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with the protocol.
* At least 18 years of age.
* Diagnosis of chronic atopic dermatitis for at least 3 years prior to enrollment.
* Subject is considered a candidate for phototherapy or systemic therapy
* Eczema Area and Severity Index (EASI) score ≥ 12
* Investigator Global Assessment (IGA) ≥ 3
* 10% body surface area (BSA) or greater
* Subject is unlikely to conceive due to male, post-menopausal, or using adequate contraceptive (barrier, hormonal, implant, or permanent sterilization methods).
* Physical exam within clinically acceptable limits.

Exclusion Criteria:

* Subject is unable to provide written informed consent or comply with the protocol.
* Subject is younger than 18 years of age.
* Subject has had atopic dermatitis for less than 3 years prior to enrollment.
* Subject with mild atopic dermatitis (EASI<12 and IGA<3) or is not a candidate for phototherapy or systemic treatments.
* Subject with current, or a history of, severe atopic dermatitis well controlled on current therapy.
* Serious known infection.
* History of immunosuppression (including human immunodeficiency virus (HIV))
* History of malignancy within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
* Severe concomitant illnesses.
* Having used immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.) or phototherapy within 4 weeks before the baseline visit.
* Treatment with topical corticosteroid or topical calcineurin inhibitor within 1 week before the baseline visit.
* Treatment with any cell-depleting agents including but not limited to rituximab: within 6 months before the baseline visit, or until lymphocyte count returns to normal, whichever is longer, or use of other biologics: within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever is longer.
* Physical or laboratory exam not within clinically acceptable limits.
* Subjects possess other diagnoses that, in the investigator's opinion, preclude him/her from safely participating in this study or interfere with the evaluation of the subject's atopic dermatitis.
* History of known or suspected intolerance to any of the ingredients of the investigational study product.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>10 mIU/mL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Liao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dupilumab Treatment: Single group study. Approximately 15 subjects will receive dupilumab for a treatment period of 52 weeks (i.e. last injection on week 50). All subjects will undergo skin biopsies for molecular profiling as well as skin and stool microbiome sampling and patch testing and different points of the study.
  Dupilumab: Dupilumab treatment
  After completion of the study, 17 were enrolled and 14 participants total completed the study.
Period: Overall Study
Arm/Group | Dupilumab Treatment
Started | 17
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Dupilumab Treatment: 14 subjects competed (3 withdrew during course of study). Subjects will received dupilumab for a treatment period of 52 weeks (i.e. last injection on week 50). All subjects will undergo skin biopsies for molecular profiling.
  Dupilumab: Dupilumab treatment
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 38.1 [21 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 17
EASI score [Mean (Full Range); unit: units on a scale] — Eczema area and severity index (EASI) is used to estimate eczema severity using 4 components: erythema, edema/papulation, lichenification, and excoriation graded from 0(none)-3(severe). Area affected is estimated in the 4 body regions separately (head/neck, upper extremities, trunk, lower extremities) and assigned an area score: 1 (1%-9%), 2 (10%-29%), 3 (30%-49%), 4 (50%-69%), 5 (70%-89%), or 6 (90%-100%). Total scores range from 0 (clear) to 72 (most severe), to be interpreted as follows:
  Almost clear: 0-1.1 Mild: 1.1-7.0 Moderate: 7.1-21.0 Severe: 21.1-50.0 Very severe: 50.0-72.0
  units on a scale | 21.98 [9 to 45.6]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in CD4+ T Effector Cells Expressing IL4 in Dupilumab-treated Subjects at Week 12 vs Week 0
Description: The percent change in CD4+ T effector cells expressing IL-4 in dupilumab-treated subjects at week 12 vs week 0 was calculated as follows. A single value was derived for the entire population with pooled samples from pre- and post-intervention time points, which was then used to calculate a percent change between the two periods. Specifically, the mean M1 across subjects of the percentage of CD4+ T effector cells expressing IL4 was computed at week 0. The mean M2 across subjects of the percentage of CD4+ T effector cells expressing IL4 was computed at week 12. The final result was calculated as: (M1-M2)/M1*100. Therefore, the result is a number and there is no central tendency metric.
Time Frame: 12 weeks
Population: Number of subjects with atopic dermatitis with single cell data
Measure: Number; unit: Percent change
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 12
Percent change
  Percent change in lesional skin | 68.4
  Percent change in non-lesional skin: number analyzed (Participants) | 6
  Percent change in non-lesional skin | 100.0

2. Secondary Outcome: Number of Differentially Expressed Genes in Cutaneous CD4+ T Cells Between Week 0 and Week 12 in Dupilumab-treated Subjects
Description: A single value was derived for the entire population with pooled samples from pre- and post-intervention time points, which was then used to calculate an percent change between the two periods. Specifically, single cell RNA-sequencing was used to calculate the number of differentially expressed genes in cutaneous CD4+ T cells between week 0 and week 12 in dupilumab-treated subjects. The calculation was performed in the software package Seurat (RRID:SCR_016341) using the FindMarkers function, which utilizes a non-parametric Wilcoxon rank-sum test. Genes were considered significantly differentially expressed if the adjusted p-value < 0.05 and the absolute value of log2(Fold Change) > 1.0. Therefore, this measure is reported as a number and there is no central tendency metric.
Time Frame: 12 weeks
Population: Number of subjects with atopic dermatitis with single cell data available
Measure: Number; unit: differentially expressed genes
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 12
differentially expressed genes
  DEG in lesional skin | 81
  DEG in non-lesional skin | 186
Statistical Analysis 1: Comparison: Dupilumab Treatment; Single cell RNA-sequencing was used to calculate the number of differentially expressed genes in cutaneous CD4+ T cells between week 0 and week 12 in dupilumab-treated subjects. The calculation was performed in the software package Seurat (RRID:SCR_016341) using the FindMarkers function, which utilizes a non-parametric Wilcoxon rank-sum test. Genes were considered significantly differentially expressed if the adjusted p-value < 0.05 and the absolute value of log2(Fold Change) > 1.0; Test type: Superiority — Note: Our statistical test was run to identify the number of significant genes. The result is a number and there is no calculation of any comparative statistic such as an odds ratio; p < 0.05, Wilcoxon (Mann-Whitney) — P-value was adjusted for false discovery rate

ADVERSE EVENTS:
Time Frame: Through study completion, up to 52 weeks.
Description: Patient reported
Arm/Group | Dupilumab Treatment
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 10/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab Treatment (N=17)
Eye irritation (Eye disorders) | 6 (8) — Patients describing dry, itchy, irritated, red, or crusty eyes. Patient reported.
Deep root cavity (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient had cavity treated and resolved with dental care
migraine (Nervous system disorders) | 1 (1)
Oral/facial herpes simplex (Infections and infestations) | 3 (4)
upper respiratory illness not otherwise defined (Infections and infestations) | 1 (1)
COVID19 (moderate) (Infections and infestations) | 1 (1)
Right ear hearing loss 2/2 Meniere's Disease (Ear and labyrinth disorders) | 1 (1)
Facial dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT03293030/Prot_SAP_000.pdf